CLINICAL TRIAL: NCT04045171
Title: Population Pharmacokinetics of Tacrolimus for Optimal Dose in Patients With Nephrotic Syndrome
Brief Title: Population Pharmacokinetics of Tacrolimus in Nephrotic Syndrome
Acronym: PISTONS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: Hunan Provincial People's Hospital (Other); ZhuZhou Central Hospital (Other); First People's Hospital of Chenzhou (Other)
Responsible Party: Sponsor
Other Study IDs: XY3-IIT-TAC1905A01
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Nephrotic Syndrome; Tacrolimus; Pharmacokinetics
Keywords: Nephrotic Syndrome; Tacrolimus; Population Pharmacokinetics
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biospecific nonspecimen specimen will be collected for the PK analysis of Tacrolimus and the gene information of Cytochrome P450 3A (CYP3A)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus, oral, 0.05-0.075 mg/kg/d, Q12h, 6～12 months

SUMMARY:
This study will use a multi-center, prospective design, with a "Real World Study" model, to include 200 patients with nephrotic syndrome. based on the Population Pharmacokinetics (PPK) model, it will study genotype and clinical factors in patients with nephrotic syndrome, to explore the Pharmacokinetics/ Pharmacodynamics (PK/PD) relationship of Tacrolimus in patients with nephrotic syndrome, and develop an optimal medication regimen.

ELIGIBILITY:
Inclusion Criteria:

* （1）Patients with Nephrotic Syndrome：

  1. Proteinuria greater than 3.5 g/24 hour
  2. Serum albumin <30 g/l
  3. Clinical evidence of peripheral oedema
  4. Hyperlipidemia 1) and 2) are necessary for diagnosis.
* （2）18-75years old（include 75），gender is not limited；
* （3）Voluntary signing informed consent。

Exclusion Criteria:

* （1）Secondary nephrotic syndrome；
* （2）Allergic to Tacrolimus or other unsuitable use of Tacrolimus；
* （3）With other immunosuppressive agents such as cyclosporin A, cyclophosphamide, mycophenolate mofetil, leflunomide, tripterygium wilfordii (hormone is not restricted)；
* （4）Severe liver dysfunction (transaminase > 3 ULN, or bilirubin > 3 ULN)；
* （5）Severe renal insufficiency（eGFR<30 ml/min/1.73m2）
* （6）Joined other clinical trials within 1 month；
* （7）Missing clinical data；
* （8）Pregnancy, lactation or planning for pregnancy within 12 months；
* （9）Researchers believe that patients who are not suitable for this clinical trial。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Nephrotic Syndrome are suit for use of Tacrolimus.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-08-10 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
change of plasma concentration of Tacrolimus | at 0hour，2hours，4hours，6hours，9hours，12hours after oral administration
  Study the plasma concentration of Tacrolimus in patients with nephrotic syndrome

SECONDARY OUTCOMES:
Genotypes as measured by next generation sequencing | one week
  Genotypes as measured by next generation sequencing

CONTACTS AND LOCATIONS:
Overall Officials: ZHIJUN HUANG, Dr., Principal Investigator — The Third Xiangya Hospital of Central South University

IPD SHARING:
Plan to Share IPD: No
We welcomes researchers interested in collaboration. We request a short research proposal including information on the background, research questions and methods, timetable and budget, and authorship. For more information please contact the principal investigator.

REFERENCES:
- [Background] Lu T, Zhu X, Xu S, Zhao M, Huang X, Wang Z, Zhao L. Dosage Optimization Based on Population Pharmacokinetic Analysis of Tacrolimus in Chinese Patients with Nephrotic Syndrome. Pharm Res. 2019 Feb 4;36(3):45. doi: 10.1007/s11095-019-2579-6. PMID 30719576
- [Background] Hao GX, Huang X, Zhang DF, Zheng Y, Shi HY, Li Y, Jacqz-Aigrain E, Zhao W. Population pharmacokinetics of tacrolimus in children with nephrotic syndrome. Br J Clin Pharmacol. 2018 Aug;84(8):1748-1756. doi: 10.1111/bcp.13605. Epub 2018 May 22. PMID 29637588
- [Background] Radhakrishnan J, Cattran DC. The KDIGO practice guideline on glomerulonephritis: reading between the (guide)lines--application to the individual patient. Kidney Int. 2012 Oct;82(8):840-56. doi: 10.1038/ki.2012.280. Epub 2012 Aug 15. PMID 22895519